CLINICAL TRIAL: NCT01596179
Title: Technology Enhanced Nurse Navigator Trial (TENN Trial) Phase III Randomized Controlled Trial
Brief Title: Technology Enhanced Nurse Navigator Trial (TENN Trial)
Acronym: TENN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mercy Medical Center (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other); Maryland Department of Health and Mental Hygiene (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MMC2011-001
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-01

CONDITIONS: Medication Adherence
Keywords: treatment adherence; fatigue; symptom management
MeSH Terms: conditions — Medication Adherence; Treatment Adherence and Compliance; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interactive navigational support (Experimental): Patients on the intervention arm are provided with a netbook computer and internet access with ongoing interaction with a nurse and a social worker navigators for a one year period.
  Interventions: Behavioral: Interactive navigational support
- control arm (Active Comparator): Patients on the control arm are provided with a netbook computer, internet access and general website information but no interactive navigational support for a one year period.
  Interventions: Behavioral: Internet access

INTERVENTIONS:
Behavioral: Interactive navigational support — Interactive navigational support is provided by a nurse and social worker navigators
  Arms: Interactive navigational support
Behavioral: Internet access — a netbook computer with internet access is provided to participants on the control arm.
  Arms: control arm

SUMMARY:
The purpose of the Technology Enhanced Nurse Navigator Trial (TENN) Trial is to find the best way to provide breast cancer patients with information through a computer connected to the internet. The study will determine if giving information during treatment may help patients cope better with their treatment. The hypothesis is that participants assigned to receive Technology-Enhanced Nurse-directed Navigation will be more likely to adhere to treatment regimens and have improved symptom management than women who have access to the education portal only.

DETAILED DESCRIPTION:
Treatment for breast cancer has been proven to decrease death from breast cancer. The key to the success of treatment is getting the right dose at the right time, but many women do not receive optimum treatment. Treatment delays, missed appointments, and failure to take medication on a regular basis lead to poorer survival from breast cancer. In a study among low income women only 60% of women adhered to the treatment, that is, taking their medication at least 80% of the time. Twenty percent of women, who were supposed to take 5 years of hormone treatment, had stopped their medication in the first year. Similar problems occur with chemotherapy and radiation therapy. Many barriers interfere with adherence to treatment, including poor symptom management, missed appointments, and cancelled appointments. Nurse navigation can help manage and minimize symptoms, assist with appointment reminders, and answer questions to obtain optimum breast cancer treatment. The goal of the proposed study is to rigorously test the delivery of nurse-navigation through a web-based knowledge and communication portal (Technology Enhanced Nurse-directed Navigation (TENN) for its impact on treatment adherence and symptom management. The success of this program will be measured by improved treatment adherence, health outcome measures such as fatigue and symptom management, patient-reported quality of life, reduced distress, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the BCCDT program for the adjuvant treatment of breast cancer,currently on medical assistance,or with an income that does not exceed 300% of the Federal Poverty Level, based on family size.
* English-speaking
* Able to give informed consent
* Not enrolled in another case-management program
* Residing within the Verizon 3G Coverage area

Exclusion Criteria:

* Non-English speaking
* Enrolled in a case management program.
* Unable to sign an informed consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Treatment Adherence | Baseline, 6 months and 12 months
  Adherence will be determined by review of the claims data. All claims, including hormone, chemotherapy and radiation therapy, doctor's visits, and hospitalizations, are sent through the BCCDT program. For chemotherapy and radiation therapy, relative dose intensity (RDI) will be measured. Adherence to hormone therapy will be measured as the medication possession ratio (MPR).A self-reported measure of adherence will be correlated with these more objective measures (Morisky et al. 1986).
Fatigue | Baseline, 6 months and 12 months
  Fatigue will be measured using a visual analogue scale. The FACT-B will be used to measure quality of life. The FACT-B is the Functional Assessment of Cancer Therapy-Breast, a reliable and valid measure for assessing subjective health-related quality of life among breast cancer survivors (Brady et al. 1997). The FACT-B includes both the FACT-General (FACT-G) and the Breast Cancer Subscale (BCS). The FACT-B has shown high internal consistency with a Cronbach's alpha of 0.90 (Brady et al. 1997).

SECONDARY OUTCOMES:
Patient satisfaction | Baseline, 6 months and 12 months
  As recommended by the NCI Navigation Research Program, we will include the Communication and Attitudinal Self-Efficacy scale for cancer (CASE-cancer) designed to measure self-efficacy and positive attitude for cancer patients (Wolf et al. 2005).
Quality of life | Baseline, 6 months and 12 months
  As a measure of distress, we will use the Impact of Events scale revised (IES-R), an updated version of the original Impact of Events scale (IES) (Horowitz et al. 1979;Weiss et al. 1997). The IES-R is a validated measure of responses to a stressful life event and addresses distress and intrusive thoughts consistent with responses to the DSM-IV diagnosis criteria of PTSD. The IES-R is readily modified to address an event such as diagnosis of cancer or a chemotherapy-related adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Helzlsouer, M.D., M.H.S., Principal Investigator — The Prevention and Research Center at Mercy Medical Center
Locations (1):
- The Prevention and Research Center at Mercy Medical Center, Baltimore, Maryland, United States